CLINICAL TRIAL: NCT04103684
Title: Low Dose Versus High Dose Steroids in Treatment of Viral Encephalitis
Brief Title: Steroids in Treatment of Viral Encephalitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AA Nagy, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LDVHDSE
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Encephalitis, Viral
MeSH Terms: conditions — Encephalitis, Viral | interventions — Methylprednisolone; Prednisolone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients will receive steroid pulse therapy (Experimental)
  Interventions: Drug: Methylprednisolone
- Patients will receive low dose steroids (Active Comparator)
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Methylprednisolone — 30mg per kg per day for 5 days followed by course of oral prednisolone
  Other Names: Prednisolone
  Arms: Patients will receive steroid pulse therapy
Drug: Dexamethasone — 0.6mg per kg perday for 5 days
  Arms: Patients will receive low dose steroids

SUMMARY:
acute viral encephalitis is used to describe restricted CNS involvement (namely, involvement of the brain, sparing the meninges)

DETAILED DESCRIPTION:
Viral encephalitis is a medical emergency The spectrum of brain involvement and the prognosis are dependent mainly on the specific pathogen and the immunological state of the host.

Although specific therapy is limited to only several viral agents, correct immediate diagnosis and introduction of symptomatic and specific therapy has a dramatic influence upon survival and reduces the extent of permanent brain injury in survivors Epidemiologic studies estimate the incidence of viral encephalitis at 3.5 to 7.4 per 100,000 persons per year. Overall, viruses are the most common cause of encephalitis.

The Centers for Disease Control and Prevention (CDC) estimates an annual incidence of approximately 20,000 new cases of encephalitis in the United States; most are mild in nature. The mortality depends largely on the etiologic agent of the encephalitis.

Herpes simplex virus (HSV) encephalitis (HSVE) is the most common cause of sporadic encephalitis in humans. More than 90% of HSVE cases are attributable to HSV type-1 (HSV-1). Approximately 5% of them are caused by HSV type-2 HSVE is a severe disease, often leading to high morbidity (40%) and mortality (up to 15% in treated cases and 70% in untreated cases) Patients with encephalitis have an altered mental status ranging from subtle deficits to complete unresponsiveness. The typical clinical presentation includes a rapid onset of fever and impaired consciousness, often accompanied by focal neurologic signs and seizures.

The current treatment of choice is the viral replication inhibitor acyclovir. Although highly effective in reducing mortality, it only results in complete recovery in one-half of patients . Steroid therapy as an adjunctive therapy in HSVE has good anti inflammatory effect. Steroid therapy has both anti inflammatory and immunosuppressive property.

The diagnosis of viral encephalitis is suspected in the context of a febrile disease accompanied by headache, altered level of consciousness, and symptoms and signs of cerebral dysfunction. These may consist of abnormalities that can be categorized into four: cognitive dysfunction (acute memory disturbances), behavioural changes (disorientation, hallucinations, psychosis, personality changes, agitation), focal neurological abnormalities (such as anosmia, dysphasia, hemiparesis, hemianopia etc.) and seizures. After the diagnosis is suspected, the approach should consist of obtaining a meticulous history and a careful general and neurological examination.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who attending Neurology unit in Assiut University Children Hospital and diagnosed as viral encephalitis.
* Age 1month : 18 year .
* Both sexes.
* Diagnosis of viral encephalitis will be confirmed by clinical picture ,investigations and exclusion of other causes of encephalopathy

Exclusion Criteria:

* Autoimmune encephalitis
* Renal failure (any patient with abnormal renal function tests will be excluded)
* Hepatic failure ( any patient with abnormal liver function tests will be excluded)
* Metabolic disorders (any patient with abnormal level of ammonia and lactate )

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Conscious level | 5 days
  Glasgow coma scale

REFERENCES:
- [Background] Hjalmarsson A, Blomqvist P, Skoldenberg B. Herpes simplex encephalitis in Sweden, 1990-2001: incidence, morbidity, and mortality. Clin Infect Dis. 2007 Oct 1;45(7):875-80. doi: 10.1086/521262. Epub 2007 Aug 24. PMID 17806053
- [Background] Steiner I, Budka H, Chaudhuri A, Koskiniemi M, Sainio K, Salonen O, Kennedy PG. Viral encephalitis: a review of diagnostic methods and guidelines for management. Eur J Neurol. 2005 May;12(5):331-43. doi: 10.1111/j.1468-1331.2005.01126.x. PMID 15804262
- [Background] Raschilas F, Wolff M, Delatour F, Chaffaut C, De Broucker T, Chevret S, Lebon P, Canton P, Rozenberg F. Outcome of and prognostic factors for herpes simplex encephalitis in adult patients: results of a multicenter study. Clin Infect Dis. 2002 Aug 1;35(3):254-60. doi: 10.1086/341405. Epub 2002 Jul 10. PMID 12115090
- [Background] Mailles A, Stahl JP; Steering Committee and Investigators Group. Infectious encephalitis in france in 2007: a national prospective study. Clin Infect Dis. 2009 Dec 15;49(12):1838-47. doi: 10.1086/648419. PMID 19929384
- [Background] McGrath N, Anderson NE, Croxson MC, Powell KF. Herpes simplex encephalitis treated with acyclovir: diagnosis and long term outcome. J Neurol Neurosurg Psychiatry. 1997 Sep;63(3):321-6. doi: 10.1136/jnnp.63.3.321. PMID 9328248
- [Background] Whitley RJ. Viral encephalitis. N Engl J Med. 1990 Jul 26;323(4):242-50. doi: 10.1056/NEJM199007263230406. No abstract available. PMID 2195341
- [Background] Gordon B, Selnes OA, Hart J Jr, Hanley DF, Whitley RJ. Long-term cognitive sequelae of acyclovir-treated herpes simplex encephalitis. Arch Neurol. 1990 Jun;47(6):646-7. doi: 10.1001/archneur.1990.00530060054017. PMID 2346392
- [Background] Tunkel AR, Glaser CA, Bloch KC, Sejvar JJ, Marra CM, Roos KL, Hartman BJ, Kaplan SL, Scheld WM, Whitley RJ; Infectious Diseases Society of America. The management of encephalitis: clinical practice guidelines by the Infectious Diseases Society of America. Clin Infect Dis. 2008 Aug 1;47(3):303-27. doi: 10.1086/589747. PMID 18582201
- [Background] Solomon T, Michael BD, Smith PE, Sanderson F, Davies NW, Hart IJ, Holland M, Easton A, Buckley C, Kneen R, Beeching NJ; National Encephalitis Guidelines Development and Stakeholder Groups. Management of suspected viral encephalitis in adults--Association of British Neurologists and British Infection Association National Guidelines. J Infect. 2012 Apr;64(4):347-73. doi: 10.1016/j.jinf.2011.11.014. Epub 2011 Nov 18. PMID 22120595
- [Background] Steiner I, Budka H, Chaudhuri A, Koskiniemi M, Sainio K, Salonen O, Kennedy PG. Viral meningoencephalitis: a review of diagnostic methods and guidelines for management. Eur J Neurol. 2010 Aug;17(8):999-e57. doi: 10.1111/j.1468-1331.2010.02970.x. Epub 2010 Mar 3. PMID 20236175
- [Background] Ramos-Estebanez C, Lizarraga KJ, Merenda A. A systematic review on the role of adjunctive corticosteroids in herpes simplex virus encephalitis: is timing critical for safety and efficacy? Antivir Ther. 2014;19(2):133-9. doi: 10.3851/IMP2683. Epub 2013 Sep 6. PMID 24009096